CLINICAL TRIAL: NCT02532751
Title: Effects of Body Contouring Surgery in Obese Patients: a Prospective Study
Brief Title: Effects of Body Contouring Surgery in Obese Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jussi Repo, MD, Helsinki University Central Hospital
Other Study IDs: 204/13/03/02/15/1
Record Dates: First submitted 2015-08-17; First posted 2015-08-26 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Validation Study; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is twofold; 1) to assess the psychometric properties of the Finnish version of the BODY-Q questionnaire, 2) to assess the effects of body contouring surgery using patient-reported outcome measures.

DETAILED DESCRIPTION:
The BODY-Q is translated into Finnish through forward and backward translation and a committee review. The preliminary version is pilot tested with 20 participants undergoing body contouring surgery.

The study is of longitudinal design gathering data from participants undergoing body contouring surgery due to obesity. Data collection takes place in the Department of Plastic Surgery, Helsinki University Central Hospital, Helsinki, Finland. The participants fill in three patient-reported outcome measures.

The outcomes of the three patient-reported outcome measures are compared with each other and internal validity assessed. Test-retest reliability is assessed after two weeks from the first completion of the questionnaires. With validated questionnaires the effects of body contouring surgery is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Body contouring surgery due to:

A) massive weight loss B) Postbariatric weight loss

* Patient age over 18 years

Exclusion Criteria:

* Patient age under 18 years
* No body contouring surgery
* Surgical intervention performed in another hospital than Helsinki and Uusimaa Hospital District
* No obesity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients who underwent body contour surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Validity of the Finnish version of the BODY-Q questionnaire | 6 months
  The psychometric properties of the BODY-Q patient-reported outcome measure are measured
Health-related quality of life after body contouring surgery in obese patients | 0.5 to 3 years
  Health-related quality of life is assessed with a questionnaire
Depression after body contouring surgery in obese patients | 0.5 to 3 years
  Depression is assessed with a questionnaire
Body image after body contouring surgery in obese patients | 0.5 to 3 years
  Body image is assessed with a questionnaire

SECONDARY OUTCOMES:
The 15-Dimensions health-related quality of life instrument | 0.5 to 3 years
  Assessment of health-related quality of life
The BODY-Q questionnaire | 0.5 to 3 years
  Assessment of health-related quality of life and body image
The Raitasalo Beck Depression Index questionnaire | 0.5 to 3 years
  Assessment of depression

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Jorvi Central Hospital, Espoo, Uusimaa
  - Helsinki University Central Hospital, Helsinki, Uusimaa